CLINICAL TRIAL: NCT02205398
Title: A Phase Ib, Open-label, Multicenter, Dose Escalation and Expansion Study, to Evaluate the Safety, Pharmacokinetics and Activity of INC280 in Combination With Cetuximab in c-MET Positive CRC and HNSCC Patients Who Have Progressed After Anti-EGFR Monoclonal Antibody Therapy.
Brief Title: Study of Safety and Efficacy of INC280 and Cetuximab, in Adult c-MET Positive mCRC and HNSCC Patients After Progression on Cetuximab or Panitumumab Therapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC280X2104; 2014-000579-20 (EudraCT Number)
Record Dates: First submitted 2014-07-25; First posted 2014-07-31 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Squamous Cell Carcinoma of Head and Neck (SCCHN); Metastatic Colorectal Cancer
Keywords: INC280; c-MET inhibitor; cetuximab; metastatic colorectal cancer; head and neck; squamous cell carcinoma; resistance to cetuximab/panitumumab; SCCHN,; cancer; oral and nasal cavity; paranasal sinuses; pharynx; larynx; parotid glands; lympth nodes of neck; mucosal lining; epithelium; colon; large intestine; rectal cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Colorectal Neoplasms; Carcinoma, Squamous Cell; Neoplasms; Laryngeal Diseases; Rectal Neoplasms | interventions — capmatinib; Cetuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- c-MET positive mCRC and HNSCC (Experimental): c-MET positive and K/NRAS WT mCRC and c-MET positive HNSCC patients
  Interventions: Drug: INC280; Drug: cetuximab

INTERVENTIONS:
Drug: INC280
Drug: cetuximab

SUMMARY:
This was an open-label, phase Ib, multicenter clinical trial to determine the MTD/RDE of the orally administered c-MET inhibitor INC280 in combination with cetuximab. This combination was to be explored in c-MET positive mCRC and HNSCC patients whose disease progressed on cetuximab or panitumumab treatment. The dose escalation part was to be guided by a Bayesian Logistic Regression Model with overdose control. At MTD/RDE, additional mCRC and HNSCC patients who progressed on cetuximab or panitumumab treatment were to be enrolled in two expansion groups to further assess the anti-tumor activity and the safety and tolerability of the combination of INC280 and cetuximab. Patients were to receive INC280 on a continuous bid dosing regimen and cetuximab every week. A treatment cycle was defined as 28 days with no scheduled break between cycles.

The trial was terminated because of difficulties in identifying patients who met the eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years
* Metastatic colorectal cancer or head and neck squamous cell carcinoma
* c-MET positive (defined by c-MET IHC intensity score +2 in ≥ 50% of tumor cells and MET gene copy number ≥ 5 by FISH or IHC intensity score +3 in ≥ 50% of tumor cells) and K/NRAS WT status for mCRC patients only
* At least one previous line of treatment for the metastatic disease and the last treatment must have included cetuximab or panitumumab. Documentation of clinical benefit and subsequent progression on cetuximab or panitumumab as the most recent line of treatment is required for patients in the expansion part
* Measurable disease as per RECIST v1.1
* ECOG performance status ≤ 2

Exclusion Criteria:

* Prior treatment with c-MET/HGF inhibitors
* History of severe reactions to cetuximab and/or panitumumab (except for G3 rash and G3 hypomagnesaemia)
* History of acute or chronic pancreatitis
* Active bleeding within 4 weeks prior to screening visit
* Symptomatic brain metastases
* Feeding tube dependence
* Not adequate hematologic, renal and hepatic function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-07-28 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-01-20 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) | during Cycle 1 and up to 4 weeks from the time of study treatment start
  To estimate the MTD and/or RDE of INC280 in combination with cetuximab in c-MET positive mCRC and HNSCC patients as measured by the incidence of DLTs in Cycle 1. A treatment cycle was defined as 28 days with no scheduled break between cycles.

SECONDARY OUTCOMES:
Frequency of Adverse Events (AEs)/Serious Adverse Events (SAEs) | During Cycle 1 Day 1 (C1D1) until treatment discontinuation for up to 2 years
  To characterize the safety and tolerability of the INC280 and cetuximab combination as measured by the frequency of AEs/SAEs in patients treated with the combination of INC280 and cetuximab
Overall Response Rate | Every 8 weeks from cycle 1, day 1 until the end of study for up to 3 years
  To assess preliminary anti-tumor activity of the INC280 and cetuximab combination as measured by Overall Response Rate in patients treated with the combination of INC280 and cetuximab. The end of study was upon completion of the survival follow-up period of the last patient treated with the combination of INC280 and cetuximab. A treatment cycle was defined as 28 days with no scheduled break between cycles.
Overall Survival | Every 12 weeks until the end of study for up to 3 years
  To assess additional clinical activity of the INC280 and cetuximab combination as measured by Overall Survival for patients in the expansion part of the study. The end of study was upon completion of the survival follow-up period of the last patient treated with the combination of INC280 and cetuximab.
Time versus plasma concentration profiles and basic PK parameters of INC280 | during the first 4 Cycles of treatment or up to 16 weeks from the time of study treatment start
  To characterize the PK profile of INC280 with cetuximab combination as measured by time versus plasma concentration profiles and basic PK parameters of INC280. A treatment cycle was defined as 28 days with no scheduled break between cycles.
Severity of Adverse Events (AEs)/Serious Adverse Events (SAEs) | From Cycle 1 Day 1 until treatment discontinuation for up to 2 years
  To characterize the safety and tolerability of the INC280 and cetuximab combination as measured by severity of AEs/SAEs in patients treated with the combination of INC280 and cetuximab
Frequency of dose treatment interruptions and reductions | From Cycle 1 Day 1 until treatment discontinuation for up to 2 years
  To characterize the safety and tolerability of the INC280 and cetuximab combination as measured by the frequency of dose interruptions and dose reductions in patients treated with the combination of INC280 and cetuximab
Progression Free Survival | Every 8 weeks from C1D1 until the end of study for up to 3 years
  To assess preliminary anti-tumor activity of the INC280 and cetuximab combination as measured by Progression Free Survival in patients treated with the combination of INC280 and cetuximab.The end of study was upon completion of the survival follow-up period of the last patient treated with the combination of INC280 and cetuximab.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- United States (3):
  - Massachusetts General Hospital Head & Neck, Boston, Massachusetts
  - Memorial Sloan Kettering MSKCC NY, New York, New York
  - University of Utah / Huntsman Cancer Institute Onc Dept, Salt Lake City, Utah
- Novartis Investigative Site, Leuven, Belgium
- Novartis Investigative Site, Toronto, Ontario, Canada
- France (2):
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Toulouse
- Germany (2):
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Würzburg
- Italy (2):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Milan, MI
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Valencia, Valencia

REFERENCES:
- [Derived] Delord JP, Argiles G, Fayette J, Wirth L, Kasper S, Siena S, Mesia R, Berardi R, Cervantes A, Dekervel J, Zhao S, Sun Y, Hao HX, Tiedt R, Vicente S, Myers A, Siu LL. A phase 1b study of the MET inhibitor capmatinib combined with cetuximab in patients with MET-positive colorectal cancer who had progressed following anti-EGFR monoclonal antibody treatment. Invest New Drugs. 2020 Dec;38(6):1774-1783. doi: 10.1007/s10637-020-00928-z. Epub 2020 May 14. PMID 32410080